CLINICAL TRIAL: NCT05379075
Title: Effects of Chen Taichi on the Physical and Psychological Health Among College Students
Brief Title: Effect of Chen Taichi on College Students' Physical and Psychological Health.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Qi Fengmeng, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Qi Fengmeng
Record Dates: First submitted 2022-04-28; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Issue; Physical Inactivity
Keywords: Mindfulness; Sleep quality; Physical fitness; college students; Taichi quan
MeSH Terms: conditions — Sedentary Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group will exercise Chen Taichi based on Relaxation guidelines, and the control group will exercise Chen Taichi with Coordination guidelines. Each parallel group has male and female separately.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Female students of Chen Taichi training based on Relaxation guidelines (Experimental): Relaxation theory is different from coordination. It only focuses on relaxing the body and mind to an extreme level. Previously, masters of Taichi described or taught it as "relax" or "let nature take its course." This explanation may lead to ignoring it since it is against intuition. Pavel explained the relaxation method as mastering muscle tension. The critical point of Pavel's book is the viewpoint of canceling the stretch reflection. The present study applied this viewpoint to judge the extent and rotation degree when practicing taichi. In other words, students will be taught this skill to relax their bodies when the tension comes out from low posture movements. The relaxation skills also include "dropping the control of the body," "exhale when stretching," "moving like a string puppet without muscle power," "steps like cats," and "three-line relaxation method." Duration:12 weeks. Frequency: 3 times per week. Time length: 90min+60min×2
  Interventions: Other: 26 styles of Chen Taichi training based on Relaxation guidelines
- Male students of Chen Taichi training based on Relaxation guidelines (Experimental): Relaxation theory is different from coordination. It only focuses on relaxing the body and mind to an extreme level. Previously, masters of Taichi described or taught it as "relax" or "let nature take its course." This explanation may lead to ignoring it since it is against intuition. Pavel explained the relaxation method as mastering muscle tension. The critical point of Pavel's book is the viewpoint of canceling the stretch reflection. The present study applied this viewpoint to judge the extent and rotation degree when practicing taichi. In other words, students will be taught this skill to relax their bodies when the tension comes out from low posture movements. The relaxation skills also include "dropping the control of the body," "exhale when stretching," "moving like a string puppet without muscle power," "steps like cats," and "three-line relaxation method." Duration:12 weeks. Frequency: 3 times per week. Time length: 90min+60min×2
  Interventions: Other: 26 styles of Chen Taichi training based on Relaxation guidelines
- Female students of Chen Taichi training based on Coordination guidelines (Active Comparator): Coordination theory is also called "three in one." It mainly guides exercisers to practice Taichi by integrating the mind, movements, and breathing in a unity state. Students in this group will be taught how to integrate the three requests according to the principles. The principles are "Waist axis," "Movements softy and slowly," "Inspiratory contraction and Expiratory stretch." The training will be conducted on the warming-up time by practicing a single movement and the club time by practicing a learned routine.
  Duration:12 weeks. Frequency: 3 times per week. Time length: 90min+60min×2
  Interventions: Other: 26 styles of Chen Taichi training based on Coordination guidelines
- Male students of Chen Taichi training based on Coordination guidelines (Active Comparator): Coordination theory is also called "three in one." It mainly guides exercisers to practice Taichi by integrating the mind, movements, and breathing in a unity state. Students in this group will be taught how to integrate the three requests according to the principles. The principles are "Waist axis," "Movements softy and slowly," "Inspiratory contraction and Expiratory stretch." The training will be conducted on the warming-up time by practicing a single movement and the club time by practicing a learned routine.
  Duration:12 weeks. Frequency: 3 times per week. Time length: 90min+60min×2
  Interventions: Other: 26 styles of Chen Taichi training based on Coordination guidelines

INTERVENTIONS:
Other: 26 styles of Chen Taichi training based on Relaxation guidelines — The arms and legs and the spine should rotate follow the arrow tips in order to cause a stretch reflex slightly. And then, the exerciser should use relaxation skills to eliminate the stretch reflex, such as exhaling, drop the control of body
  Arms: Female students of Chen Taichi training based on Relaxation guidelines; Male students of Chen Taichi training based on Relaxation guidelines
Other: 26 styles of Chen Taichi training based on Coordination guidelines — When the posture needs to open the arms should accompany with "inhale" and when the posture needs to close the arms should accompany with "exhale". Similarly, if the arm is lifting should accompany with inhale, and the put down should accompany with exhale.
  Arms: Female students of Chen Taichi training based on Coordination guidelines; Male students of Chen Taichi training based on Coordination guidelines

SUMMARY:
Tai Chi is a kind of traditional martial arts in China, which has a remarkable function in healthcare. It has been used in many diseases as a complementary theory. The Chinese government attaches much importance to university students' physical and psychological health. However, there is an indisputable fact that the health condition of university students is declining, according to the report of the education ministry of China 2021. Tai Chi is a solid supplement to physical education and how to improve the physical health of university students through Tai Chi is the key to university physical education. This experimental research examines the effectiveness and the differences of two types of Chen Taichi training methods on the physical and psychological health of college students in China. Finally, to evaluate if the Chen Taichi with developed guidelines can improve the college students' physical and psychological health.

DETAILED DESCRIPTION:
The research is a two-group randomized control experiment. The control group (CG) will accept the training of Chen Taichi under the guideline of the "three in one" theory which means the integration of slow circular movements, breath regulation, and concentration or mindfulness. The experimental group (EG) will practice Chen Taichi under relaxation theory which combines the "Body-rotation" and "Relax into Stretch". all other conditions will be kept as same as possible, such as the Chen Taichi routine.

An example of one Chen Taichi posture of EG. The arms and legs and the spine should rotate follow the arrow tips in order to cause a stretch reflex slightly. And then, the exerciser should use relaxation skills to eliminate the stretch reflex, such as exhaling, and drop the control of the body. Relax into Stretch: Instant flexibility through mastering muscle tension. The body-rotation levels should be added in steps with the process of practice. It does not need to accompany breathing except the relaxation needs to exhale. Most of the time breathing is common daily.

Content of Chen Taichi movements:

1、Preparing form 2、Buddha's Warrior attendant pounds mortar 3、Lazy about tying coat 4、Six sealing and four closing 5、Single whip 6、The white crane spreads its wings 7、Walk obliquely 8、Holding up the knee 9、The fist Cover Fist and Punch.

10、Buddha's Warrior attendant pounds mortar secondly. 11、Lean with back 12、Push both hands 13、The punch at the elbow's bottom 14、Step back and whirl arms on both sides 15、Turning back with arms twining 16、The second Cover Fist and Punch 17、Six sealing and four closings （secondly）18、Single whip（secondly）19、Wave hands 20、The dragon on the ground 21、Step forward with seven stars 22、Step back and mount the tiger 23、Double wave lotus 24、 The cannon right overhead 25、 Buddha's Warrior attendant pounds mortar thirdly 26、Closing form。

ELIGIBILITY:
Inclusion Criteria:

* Males and females are college students;
* Able to finish the physical fitness test;
* Without any disease of organs;
* Age ranged from 18-30;
* Not engaged in long term exercising Taichi and other Taichi derived movements.

Exclusion Criteria:

* Detained and Repeated students;
* Not willing to join the research or not willing to spend club time to train;
* Disabled students;
* Involvement in other physical activity studies such as basketball matches and so on;
* Contraindications to physical activity;
* Students good at tai chi especially once studied in kids.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change form baseline Blood pressure at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter belongs to Cardiopulmonary function.
Change form baseline Lung capacity at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter belongs to Cardiopulmonary function.
Change form baseline Rest-Heart rate at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter belongs to Cardiopulmonary function.
Change form baseline Step index at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter belongs to Cardiopulmonary function.
Change form baseline Sit-reach at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter can represent flexibility of students.
Change form baseline Shoulder-rotation at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  The parameter can represent flexibility of shoulder.
Change form baseline Body-rotation at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  The parameter can represent flexibility of spine.
Change form baseline 50m at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter represent speed of students.
Change form baseline lateral jump at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  The parameter represents speed.
Change form baseline hand-grip at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  The parameter represents power.
Change form baseline standing-leap at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  The parameter represents power.
Change form baseline enduracne runing at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Male students test 2400 meters, and female test 2000 meters.
Change form baseline Push-up at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  The parameter represents endurance of arms.
Change form baseline sit-ups at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  The parameter represenst muscluar endrance of abdominal muscle.
Change form baseline body-fat at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter represent body composition.
Change form baseline Waist-Hip Ratio at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  This parameter represents body-shape.
Change form baseline mindfulness at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Tested by the Five facet mindfulness questionnaire.It is a 39-item and five-point Likert scale instrument. This instrument developed five factors representing mindfulness elements: observing to sensation, describing these internal experiences with words, acting with awareness rather than no "automatic pilot," nonjudging of inner experiences, and nonreactivity to inner experience. The total mindfulness score is calculated by adding all scores of the five factors. Higher scores mark higher levels of mindfulness.
Change form baseline Mood at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Tested by The Profile of Mood State.The POMS is a brief measure of 7 dimensions of dispositional mood that can discriminate among individuals at both positive and negative mood construct. It is a five-point Likert format questionnaire (1=not at all, 5=extremely) that involves a 40-item adjective. The 40-item includes nervousness, anger, tiredness, depression, energy, panic, and self-esteem. Energy and self-esteem represent the upbeat mood, and the other four express the negative mood. The total score is calculated by subtracting the total negative score from the total positive score.
Change form baseline Sleep quality at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Tested by The Pittsburgh Sleep Quality Index. The PSQI consists of 19 self-rated questions and five questions rated by the bed partner or roommate. The latter five questions only collect the clinical information, are not tabulated in the scoring of the PSQI. The 19 self-rated questions assess a wide variety of factors relating to sleep quality, including estimates of sleep duration and latency and of the frequency and severity of specific sleep-related problems. These 19 items are categorized into seven component scores, each weighted equally on a 0-3 scale. The seven component scores are then summed to yield a global PSQI score, ranging from 0-21; higher scores indicate worse sleep quality.
Change form baseline Negative emotions at 6 weeks and 12 weeks. | Pretest: Before experiment; Mid-test: 6 weeks end; Post-test: 12 weeks end.
  Tested by Depression Anxiety Stress Scales-21.This scale consists of 21 items that are rated on a four-point Likert scale ranging from 0 to 3 ("Did not apply to me at all" to "Applied to me very much or most of the time"). The items comprise three subscales: depression, anxiety, and stress. The depression subscale indicates: 0-9 are standard, 10-13 are mild, 14-20 are moderate, more than 21 are severe. The anxiety subscale rates 0-7 as usual, 8-9 as soft, 10-14 as moderate, 15-19 as severe, and 20 or higher as extremely severe. Pairwise, the stress subscale categories 0-14 as usual, 15-18 as mild, 19-25 as moderate, 26-33 as severe, and 34 or higher as extremely severe.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Fengmeng, Principal Investigator — University Putra Malaysia
Locations (1):
- Sports Human Science Laboratory, Jiaozuo, Henan, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Background] Zheng G, Lan X, Li M, Ling K, Lin H, Chen L, Tao J, Li J, Zheng X, Chen B, Fang Q. Effectiveness of Tai Chi on Physical and Psychological Health of College Students: Results of a Randomized Controlled Trial. PLoS One. 2015 Jul 6;10(7):e0132605. doi: 10.1371/journal.pone.0132605. eCollection 2015. PMID 26147842
- [Background] Caldwell K, Harrison M, Adams M, Quin RH, Greeson J. Developing mindfulness in college students through movement-based courses: effects on self-regulatory self-efficacy, mood, stress, and sleep quality. J Am Coll Health. 2010 Mar-Apr;58(5):433-42. doi: 10.1080/07448480903540481. PMID 20304755
- [Background] Nedeljkovic M, Ausfeld-Hafter B, Streitberger K, Seiler R, Wirtz PH. Taiji practice attenuates psychobiological stress reactivity--a randomized controlled trial in healthy subjects. Psychoneuroendocrinology. 2012 Aug;37(8):1171-80. doi: 10.1016/j.psyneuen.2011.12.007. Epub 2012 Jan 4. PMID 22222120
- See also: This article is from National Library of Medinice — http://pubmed.ncbi.nlm.nih.gov/22222120/
- See also: This article is from National Library of Medinice — https://pubmed.ncbi.nlm.nih.gov/20304755/
- See also: This article is from National Library of Medinice — https://pubmed.ncbi.nlm.nih.gov/26147842/